CLINICAL TRIAL: NCT05099874
Title: Feasibility and Efficacy of Attentional-Control Training in Sickle Cell Disease
Acronym: ACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Steven J. Hardy, Associate Professor of Psychiatry and Behavioral Sciences, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00016536
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease; Attention Deficit; Cognitive Deficit in Attention
MeSH Terms: conditions — Anemia, Sickle Cell; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- EndeavorRx (Experimental): Children will be asked to begin attentional control training at home within two weeks of baseline testing and to complete 6 training missions per day (25-30 minutes), 5 days per week, for 4 weeks (total = 120 training missions).
  Interventions: Device: EndeavorRx

INTERVENTIONS:
Device: EndeavorRx — EndeavorRx is a digital intervention delivered through an action video game that is indicated to improve attention function. EndeavorRx users first complete two discrete tasks: 1) a perceptual discrimination/attention task in which users respond to target stimuli and ignore distractor stimuli (e.g., tapping the screen quickly only when red aliens appear) and 2) a sensorimotor navigation task in which users tilt their device to steer a hovercraft down a river while targeting or avoiding certain objects. Users are subsequently presented with a multitask training session where they complete the perceptual discrimination/attention task and the sensorimotor navigation task simultaneously. Algorithms adapt the program in both real-time and between sessions to automatically adjust the difficulty level.

SUMMARY:
Children with sickle cell disease (SCD) exhibit significantly reduced cognitive functioning (often difficulties with attention) compared to peers and siblings without SCD. EndeavorRx (Akili Interactive Labs: Boston, MA) is an FDA-approved home-based, electronic attentional-control training program designed to treat attention problems in youth. Users access EndeavorRx on a tablet device for 25-30 minutes each day, 5 days per week, for 4 weeks. The program involves training in a game-like environment that repeatedly challenges attentional-control abilities and adapts to user performance, becoming more difficult over time as performance improves. This pilot study is examining the feasibility, acceptability, and preliminary efficacy of EndeavorRx in a sample of 20 children with SCD ages 8-16 who are being treated with chronic blood transfusion therapy.

DETAILED DESCRIPTION:
Children with sickle cell disease (SCD) exhibit significantly reduced cognitive functioning compared to peers and siblings without SCD. Cognitive deficits are greatest among those with severe SCD genotypes, persistent anemia, and strokes and these deficits worsen over time. These deficits often manifest as difficulties with executive functioning and attention due to the predominance of cerebral infarcts (>90%) that occur in the frontal cortex. Reduced capacity to engage such cognitive skills has significant real-world implications, leading to disruption to academic achievement and attainment, vocational outcomes, and quality of life. EndeavorRx (Akili Interactive Labs: Boston, MA) is an FDA-approved home-based, electronic attentional-control training program designed to treat attention problems in youth. Users access EndeavorRx on a tablet device for 25-30 minutes each day, 5 days per week, for 4 weeks. The program involves training in a game-like environment that repeatedly challenges attentional-control abilities and adapts to user performance, becoming more difficult over time as performance improves. Data support effects of EndeavorRx on performance-based and parent-reported measures of attention in youth with Attention-Deficit/Hyperactivity Disorder (ADHD). Given the similarities in attentional functioning among youth with ADHD and those with SCD, EndeavorRx holds promise as an intervention for patients experiencing SCD-related cognitive deficits. This pilot study is examining the feasibility, acceptability, and preliminary efficacy of EndeavorRx in a sample of 20 children with SCD ages 8-16 who are being treated with chronic blood transfusion therapy due to an identified high risk of stroke or as a preventive measure to protect against additional stroke events.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of SCD
* ages 8-16 years
* maintained on monthly blood transfusions consistently for at least 3 months.
* patients will be proceed to the intervention phase only if they have a T-score > 75th percentile for Omission Errors on the Conners' Continuous Performance Test, 3rd Edition (CPT-3) or a T-score > 75th percentile for the Inattention subscale of the ADHD Rating Scale, Fifth Edition (ADHD-RS-V).

Exclusion Criteria:

* estimated Intelligence Quotient < 70
* motor, visual, or auditory impairment that prevents computer use
* known diagnosis of a mental health condition that precludes, or takes treatment precedence over, participation in cognitive training
* history of photosensitive seizures
* insufficient English fluency.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
EndeavorRx feasibility assessed by patient/family interest | Approximately 10 months
  Feasibility will be determined by examining the proportion of eligible patients/families approached about the study who enroll.
EndeavorRx feasibility assessed by program completion rates | Approximately 4 weeks per participant
  Feasibility will be evaluated by examining the proportion of the sample that completes at least 60 EndeavorRx missions (50%).
EndeavorRx feasibility assessed by reports of technical ease-of-use and satisfaction | Approximately 4 weeks from start of intervention
  Feasibility will be determined by examining parent and child reports of technical ease-of-use and satisfaction.

SECONDARY OUTCOMES:
Inattention assessed by change in Omission Errors on the Conners' Continuous Performance Test, 3rd Edition (CPT-3) | Approximately 4 weeks from start of intervention
  EndeavorRx efficacy will be evaluated by examining change in Omission Errors on the CPT-3 computerized assessment after completing EndeavorRx.
Inattention assessed by change in the Inattention subscale of the ADHD Rating Scale, Fifth Edition (ADHD-RS-V) | Approximately 4 weeks from start of intervention
  EndeavorRx efficacy will be evaluated by examining change in the Inattention subscale of the parent-reported ADHD-RS-V after completing EndeavorRx.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Hardy, Ph.D., Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No